CLINICAL TRIAL: NCT07057947
Title: Is Pericapsular Nerve Group (PENG) Block Superior to Interscalene Nerve Block Regarding Motor Power Affection in Shoulder Scope Surgeries? A Randomised Comparative Study.
Brief Title: Is Pericapsular Nerve Group Block Better Than Interscalene Nerve Block Regarding Effect on Hand Movement in Shoulder Scope Surgeries?
Acronym: PENG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherin Refaat (Other)
Responsible Party: Sponsor-Investigator, Sherin Refaat, Dr. Sherine Refaat Mahmoud, Assistant Professor of anesthesiology, surgical ICU and pain management, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-323-2024
Record Dates: First submitted 2025-03-11; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Arthroscopic Surgery
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group P (Active Comparator): This arm will receive PENG block
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block; Device: Acuson X300 ultrasound,Siemens medical solution INC, Germany
- Group I (Active Comparator): This arm will receive interscalene block
  Interventions: Procedure: Interscalene Nerve Block; Device: Acuson X300 ultrasound,Siemens medical solution INC, Germany

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — Injection of local anesthetic between deltoid muscle and subcapsularis tendon
  Arms: Group P
Procedure: Interscalene Nerve Block — Injection of local anesthetic between anterior and middle scalene muscles around the roots of brachial plexus
  Arms: Group I
Device: Acuson X300 ultrasound,Siemens medical solution INC, Germany — high frequency linear probe

SUMMARY:
The goal of this clinical trial is to learn if pericapsular nerve group block (PENG) in shoulder scope surgery provides adequate analgesia with less affection of muscle power compared to interscalene block. The main questions it aims to answer are:

Does PENG block provide analgesia similar to interscalene block? Does PENG block have less or no effect on muscle power compared to interscalene block? Researchers will compare PENG block with interscalene block

Participants will:

Receive either PENG or interscalene block before shoulder scope surgery Be evaluated for their motor power after receiving the block and after the surgery Be evaluated for pain after the surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of the specified age range
* Any gender
* American Society of Anaesthesiologists physical status grades 1 and 2
* Body mass index less than 35
* Duration of surgery between 90 to 120 minutes

Exclusion Criteria:

* American Society of Anaesthesiologists physical status grades 3 and 4
* Allergy to local anesthetics
* Coagulation disorder (INR >1.2, Platelets <100,000), or recent intake of clopidogrel or warfarin within 1 week
* Active infection at site of injection

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time for full recovery of hand motor power | Starting from block activation until the achieves preoperative grip strength ( 24 hours)
  Time from start of block activation till time of achieving grip strength similar to patient's baseline

SECONDARY OUTCOMES:
Hand grip power after surgery | 2,4,6,12,24 hours
  The measured hand grip power using a digital dynamometer
Visual analogue scale assessment | 2,4,6,12 hours
  Assessing postoperative pain, scale from 0 to 10 where 0 is no pain and 10 is worst pain
Time to first analgesia request | 24 hours
  Time from end of the surgery till the participant asks for additional analgesia
Patient satisfaction score | 24 hours
  Assessing the participant satisfaction after the postoperative period regarding overall experience with the block given on a scale of 1 to 5, where 1 is the least satisfaction and 5 is the greatest.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Mosaffa F, Taheri M, Manafi Rasi A, Samadpour H, Memary E, Mirkheshti A. Comparison of pericapsular nerve group (PENG) block with fascia iliaca compartment block (FICB) for pain control in hip fractures: A double-blind prospective randomized controlled clinical trial. Orthop Traumatol Surg Res. 2022 Feb;108(1):103135. doi: 10.1016/j.otsr.2021.103135. Epub 2021 Oct 29. PMID 34715388
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Background] Hussain N, Goldar G, Ragina N, Banfield L, Laffey JG, Abdallah FW. Suprascapular and Interscalene Nerve Block for Shoulder Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2017 Dec;127(6):998-1013. doi: 10.1097/ALN.0000000000001894. PMID 28968280
- [Background] Stasiowski M, Zuber M, Marciniak R, Kolny M, Chabierska E, Jalowiecki P, Pluta A, Missir A. Risk factors for the development of Horner's syndrome following interscalene brachial plexus block using ropivacaine for shoulder arthroscopy: a randomised trial. Anaesthesiol Intensive Ther. 2018;50(3):215-220. doi: 10.5603/AIT.a2018.0013. Epub 2018 Jun 22. PMID 29931665
- [Background] Bergmann L, Martini S, Kesselmeier M, Armbruster W, Notheisen T, Adamzik M, Eichholz R. Phrenic nerve block caused by interscalene brachial plexus block: breathing effects of different sites of injection. BMC Anesthesiol. 2016 Jul 29;16(1):45. doi: 10.1186/s12871-016-0218-x. PMID 27473162
- [Background] Paul RW, Szukics PF, Brutico J, Tjoumakaris FP, Freedman KB. Postoperative Multimodal Pain Management and Opioid Consumption in Arthroscopy Clinical Trials: A Systematic Review. Arthrosc Sports Med Rehabil. 2021 Dec 17;4(2):e721-e746. doi: 10.1016/j.asmr.2021.09.011. eCollection 2022 Apr. PMID 35494281
- [Background] Guity MR, Sobhani Eraghi A, Hosseini-Baharanchi FS. Early postoperative pain as a risk factor of shoulder stiffness after arthroscopic rotator cuff repair. J Orthop Traumatol. 2021 Jun 26;22(1):25. doi: 10.1186/s10195-021-00585-9. PMID 34173872
- [Background] Calvo E, Torres MD, Morcillo D, Leal V. Rotator cuff repair is more painful than other arthroscopic shoulder procedures. Arch Orthop Trauma Surg. 2019 May;139(5):669-674. doi: 10.1007/s00402-018-3100-0. Epub 2018 Dec 17. PMID 30560289
- [Background] Zong LZ, Duan MM, Yuan WW, Lu HD. Efficacy of shoulder arthroscopic surgery for the treatment of rotator cuff injury: A protocol of systematic review and meta-analysis. Medicine (Baltimore). 2020 Jun 26;99(26):e20591. doi: 10.1097/MD.0000000000020591. PMID 32590734
- [Background] Farmer KW, Wright TW. Shoulder arthroscopy: the basics. J Hand Surg Am. 2015 Apr;40(4):817-21. doi: 10.1016/j.jhsa.2015.01.002. Epub 2015 Feb 26. PMID 25726045

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT07057947/Prot_SAP_000.pdf